CLINICAL TRIAL: NCT02384655
Title: Effect of Fenugreek Use in Mothers of Preterm on Breast Milk Production and Macronutrient Content
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0652-14-TLV-RM
Record Dates: First submitted 2015-02-24; First posted 2015-03-10 (Estimated); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Preterms; Lactation
Keywords: Preterms; Breastfeeding; Lactation; Macronutrients
MeSH Terms: conditions — Breast Feeding | interventions — fenugreek seed meal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fenugreek (Experimental): Mothers will take fenugreek for 14 days
  Interventions: Drug: Fenugreek seed meal

INTERVENTIONS:
Drug: Fenugreek seed meal — 3x3 capsules of fenugreek seeds per day for 14 days

SUMMARY:
Feeding human milk to preterm infants does reduce the risk of serious and costly neonatal intensive care unit acquired morbidity such as NEC and the late onset sepsis.

It is often difficult to obtain sufficient quantities of human milk from mothers of preterm infants most of whom are breast pump-dependent for weeks or months. Mothers will try to use galactogogues in an attempt to increase milk production. Fenugreek (Trigonella foenum-graecum) seeds is the most commonly used herbal galactogogue and is a member of the pea family. Our experience at the NICU is that around 30% of preterm mothers desperately looking for ways to increase their breast milk supply will eventually took fenugreek (Hilbe) as food supplement. Although widely recommended, there is limited evidence to support the effectiveness of fenugreek as a galactogogue.

The aims of this study are to evaluate whether maternal consumption of fenugreek seeds has any effect on macronutrients composition of breast milk and whether fenugreek is transferred to the infant via mother milk. In addition any changes in mother and infant health status will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy mothers 7 to 14 days postpartum,
* Mothers of preterm infants under 38 weeks of gestation,
* Mothers with poor milk supply documented by professional lactation consultants.

Exclusion Criteria:

* Mothers with mastitis,
* Mothers with breast engorgement,
* Mothers currently consuming Reglan, Domperidone or other drugs/herbals used to induce milk production,
* Mothers who are taking medications (Diuretics, Pseudoephedrine, - Anticholinergics, Warfarin or any anticoagulant, An estrogen-containing birth control pill),
* Mothers with Diabetes mellitus,
* Mothers who have had breast surgery that could alter milk synthesis or production,
* Mothers diagnosed with Polycystic Ovary Syndrome,
* Mothers diagnosed with Asthma or atopic disease,
* Mothers who are known to be allergic to peanuts or soybeans,
* Mothers whose milk supply per 24 hours exceeds 600 mL,
* Mothers with hypo/hyperthyroidism

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-03-11 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change in daily volume of expressed milk | at day 0, 3, 7, 10, 14

SECONDARY OUTCOMES:
Change in Macronutrient content analysis of breastmilk | at day 0, 3, 7, 14

CONTACTS AND LOCATIONS:
Overall Officials: Ronella Marom, MD, Principal Investigator — Department of Neonatology, Lis Maternity Hospital, Tel Aviv Medical Center
Locations (1):
- Department of Neonatology Tel Aviv Medical Center, Tel Aviv, Israel